CLINICAL TRIAL: NCT00630669
Title: Randomized Study Of Endoscopic Band Ligation Versus Bipolar Probe Electrocoagulation Of Bleeding Internal Hemorrhoids
Brief Title: Comparison Between Two Endoscopic Treatments of Bleeding Internal Hemorrhoids:Band Ligation and Electrocoagulation Probe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other)
Responsible Party: Rome Jutabha,MD/Associate Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 97-10-009-03
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Last update posted 2008-03-07 (Estimated); Status verified 2001-05

CONDITIONS: Hemorrhoids
Keywords: Internal hemorrhoids; Rubber band ligation; Bipolar coagulation
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rubber band ligation
  Interventions: Procedure: Rubber band ligation
- 2 (Active Comparator): Bipolar coagulation
  Interventions: Procedure: Bipolar coagulation

INTERVENTIONS:
Procedure: Rubber band ligation — placing rubber bands around the internal hemorrhoids
  Arms: 1
Procedure: Bipolar coagulation — using electricity to cauterize
  Arms: 2

SUMMARY:
The purpose of this study is to determine which treatment, band ligation (placing rubber bands around the hemorrhoids) or BICAP electrocoagulation (using electricity to cauterize) is safer and more effective endoscopic treatment for bleeding internal hemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

1. Grade II or III internal hemorrhoids with chronic rectal bleeding, which failed at least 8 weeks of intensive medical therapy.
2. Age over 18 years
3. A life expectancy of at least 24 months
4. A signed written informed consent

Exclusion Criteria:

1. The patient was uncooperative or could not return for routine outpatient follow-up
2. Severe or end-stage co-morbid illness
3. Prior endoscopic or surgical treatment of hemorrhoids within the past 6 months
4. Ongoing need for anticoagulation therapy or high doses of aspirin or non-steroidal antiinflammatory agents
5. Presence of severe rectal pain
6. Recently thrombosed internal or external hemorrhoids
7. Anal stricture,fissure, fistula,or abscess
8. Rectal carcinoma or bleeding distal colonic polyp
9. Rectal varices
10. Acute or chronic colitis
11. Rectal prolapse
12. Radiation telangiectasia of the rectum
13. Prothrombin time >3 seconds over control
14. Platelet count <75,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1997-12; Primary Completion 2000-05 (Actual); Study Completion 2001-05 (Actual)

PRIMARY OUTCOMES:
treatment success rate | one year

SECONDARY OUTCOMES:
treatment complication rate | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Rome Jutabha,MD, Los Angeles, California, United States